CLINICAL TRIAL: NCT07075978
Title: MHWP Remote Health Study
Brief Title: The Mobile Health and Wellness Program Remote Health Study
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Principal Investigator, Lana Sargent, Associate Dean for Practice and Community Engagement, Virginia Commonwealth University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: VCU HM20031925; 1 (Other: Mobile Health and Wellness Program)
Record Dates: First submitted 2025-07-10; First posted 2025-07-20 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Diabetes Mellitus Self Management Education; Hypertension Self-management; Self Management
Keywords: Older adults; Remote patient monitoring; Telehealth; Interprofessional
MeSH Terms: interventions — Remote Patient Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telehealth (Active Comparator): This usual care group will engage with Mobile Health and Wellness Program through standard telephone visits.
  Interventions: Behavioral: Telephone
- Remote group (Experimental): This experimental remote group will engage with Mobile Health and Wellness program using remote patient monitoring devices.
  Interventions: Behavioral: Remote patient monitoring

INTERVENTIONS:
Behavioral: Remote patient monitoring — The usual interprofessional program activities are delivered via remote patient monitoring kits. The kit includes a tablet for virtual visits with the Mobile Health and Wellness Team and access to educational videos, as well as at-home monitoring devices for blood pressure, blood sugar if diabetic, pulse ox if COPD, and/or weight scale.
  Arms: Remote group
Behavioral: Telephone — The usual interprofessional program activities are delivered via telephone visits without any at-home monitoring devices.
  Arms: Telehealth

SUMMARY:
This clinical trial trial design will be a pretest-posttest comparison group pilot study that evaluates the implementation of team-based telemedicine visits and remote patient monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Participant in the Mobile Health and Wellness Program
* 18 years old or over
* Reporting with hypertension, diabetes, congestive heart failure, or chronic obstructive pulmonary disease
* English-speaking
* Currently taking blood pressure and/or diabetes medications
* Capable of engaging with the Health Recovery Solutions (HRS) Remote Patient Monitoring (RPM) device or participating in standard telephone-based care.

Exclusion Criteria:

* Prior diagnosis of Dementia; Alzheimer's disease, Lewy body, Parkinson's, or vascular dementia.
* No access to an internet connection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-17 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
PROMIS Self-Efficacy for Managing Chronic Conditions | Baseline, 8 weeks and through the end of participation at 16 weeks
  Change in self-efficacy in managing chronic conditions at 16 weeks, the tool will be the PROMIS Self-Efficacy for Managing Chronic Conditions - The PROMIS Self-Efficacy scoring system is designed to assess the confidence of individuals in managing their health and daily activities. It is based on a T-score metric, where a score of 10 points corresponds to one standard deviation (SD) from the mean. The PROMIS scoring system has a mean of 50 and a standard deviation (SD) of 10 in the US General Population. A score of 40 is one SD lower than the mean, while a score of 60 is one SD higher. This scoring system is used to evaluate the self-efficacy for managing chronic conditions and daily activities, providing a standardized way to measure and compare the effectiveness of interventions and treatments.
The Medical Outcomes Study (MOS) Measures of Patient Adherence | Baseline, 8 weeks and through the end of participation at 16 weeks
  Improved adherence to medical recommendations at 16 weeks, the tool will be The Medical Outcomes Study (MOS) Measures of Patient Adherence is a 5-item scale to assess the adherence of patients with chronic conditions to medical recommendations. To score a Medical Outcomes Study (MOS) survey, you first need to recode the raw survey responses according to the specific scale's rules. Then, you average the recoded item scores to get a subscale score. For an overall index, you average the scores for all relevant items. Finally, you can transform these average scores to a 0-100 scale, where 100 represents the best possible score.
The REALM Health Literacy | Baseline, 8 weeks and through the end of participation at 16 weeks
  Change in health literacy at 16 weeks, The REALM Health Literacy - Short Form is a 7-item assessment tool that is a validated rapid measure of health literacy. It is a 7-item word recognition test to screen a patient's health literacy quickly. The patient is asked to read the words aloud. Scores are interpreted into a reading grade level equivalent, takes about one minute and requires minimal training.
Change in mobile device proficiency at 16 weeks | Baseline, 8 weeks and through the end of participation at 16 weeks
  The Mobile Device Proficiency (MDPQ-16) is a 16-item survey measuring participants' ability to operate a mobile device. First, assign a numerical value from 1 to 5 to each item, with one being "Never Tried" and five being "Very Easily". Next, calculate the average score for each of the eight subscales (Mobile Device Basics, Communication, Data and File Storage, Internet, Calendar, Entertainment, Privacy, and Troubleshooting/Software Management). Finally, add the eight subscale averages to obtain a total score ranging from 8 to 40.

SECONDARY OUTCOMES:
Change in blood pressure | Baseline, 8 weeks and through the end of participation at 16 weeks
  Change in blood pressure (SBP/DBP) over the course of the 16 weeks, particularly for baseline to post-study in the remote group. Blood pressure is measured in units of millimeters of mercury (mmHg). The readings are always given in pairs, with the upper (systolic) value first, followed by the lower (diastolic) value.
Change in weight | Baseline, 8 weeks and through the end of participation at 16 weeks
  Change in weight over the course of the 16 weeks, particularly for baseline to post study in the remote group.
Change in blood oxygenation | Baseline, 8 weeks and through the end of participation at 16 weeks
  Measured by a pulse oximeter over the course of the 16 weeks, particularly for baseline to post-study in the remote group. (No range outcome necessary- continuous value)
Change in blood glucose | Baseline, 8 weeks and through the end of participation at 16 weeks
  Change in blood glucose over the course of the 16 weeks, particularly for baseline to post study in the remote group.

CONTACTS AND LOCATIONS:
Overall Officials: Lana Sargent, Principal Investigator — Virginia Commonwealth University
Locations (1):
- School of Nursing Mobile Health and Wellness Program, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No